CLINICAL TRIAL: NCT05118633
Title: Technology Assisted Treatment for Trichotillomania
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HabitAware Inc. (Industry)
Collaborators: Kent State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R44MH114773 (NIH)
Record Dates: First submitted 2021-11-02; First posted 2021-11-12 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Trichotillomania
Keywords: Hair Pulling Disorder; Body-Focused Repetitive Behaviors; Trichotillomania
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group - HabitAware condition (Experimental): This group will receive the device which alerts the participant when performing hair pulling behavior and the app which provides psychoeducation and components of Habit Reversal Training.
  Interventions: Behavioral: Device and app system designed for participant to self-administer Habit Reversal Training and Stimulus Control
- Control group - reminder bracelet condition (Placebo Comparator): This group will receive only a device that vibrates randomly several times per hour as a reminder not to pull, as well as being asked to journal about their daily activities in an app.
  Interventions: Behavioral: Reminder bracelet and journaling app control condition

INTERVENTIONS:
Behavioral: Device and app system designed for participant to self-administer Habit Reversal Training and Stimulus Control — Participants will receive an awareness bracelet and an app that work together to implement key features of Habit Reversal Training and Stimulus Control. The participant will take part in psychoeducation, awareness training, and competing response training related to trichotillomania, as well as receive stimulus control reminders.
  Arms: Experimental group - HabitAware condition
Behavioral: Reminder bracelet and journaling app control condition — Participants will receive a bracelet programmed to vibrate randomly several times per hour during waking hours. They will be instructed this is a reminder not to pull. They will also be instructed to journal in an app on their phone several times per day.
  Arms: Control group - reminder bracelet condition

SUMMARY:
Trichotillomania is characterized by recurrent hair pulling resulting in hair loss causing significant distress and impairment which persists despite repeated attempts to stop. Behavioral based therapies focused on increasing awareness of hair pulling followed by the use of an incompatible behavior have proven effective. In an effort to enhance awareness, a wrist worn motion detection device and a companion mobile application was created. In this study, we will test the initial efficacy of the HabitAware device and accompanying app as a system for delivering self-administered habit reversal training (HRT).

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate;
* Current diagnosis of TTM (as assessed via TDI);
* Regular access to a smartphone with GPS capabilities (i.e., available for completing assessment probes throughout the day);

Exclusion Criteria:

* Currently receiving psychotherapy
* Other psychiatric condition requiring more immediate care
* Have previously used any behavior awareness devices (e.g. Keen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in clinical symptoms amongst participants | Eight weeks
  Demonstrated improvement in clinical symptoms on the MGH-HPS and/or NIMH-TSS for those in the HabitAware condition.